CLINICAL TRIAL: NCT03513822
Title: Ketamine's Efficiency in the Treatment of Chronic Pain With an Added Inflammatory Component Exploring the Kynurenin Pathway. A Randomized, Double Blind, Placebo-controlled Trial
Brief Title: Ketamine's Efficiency in the Treatment of Chronic Pain: Kynurenin Pathway
Acronym: KEKU1
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Redar (Other)
Collaborators: Hôpital Raymond Poincaré (Other); Hopital Lariboisière (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Fondation Apicil (Other); Hospital Ambroise Paré Paris (Other); Recherche Clinique Paris Descartes Necker Cochin Sainte Anne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REDAR; 2017-003930-10 (EudraCT Number); protocole ph-03-2018 (Registry Identifier: CPP ILE DE FRANCE X)
Record Dates: First submitted 2018-03-23; First posted 2018-05-02 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Neuralgia; Chronic Pain; Inflammation
Keywords: KETAMINE; CHRONIC PAIN; NEUROPATHIC PAIN; KYNURENINE; KYNURENINE PATHWAY; BEDSORES; ANTI-INFLAMMATORY; ULCER PRESSURE
MeSH Terms: conditions — Neuralgia; Chronic Pain; Inflammation; Pressure Ulcer | interventions — Ketamine; Midazolam

STUDY DESIGN:
Intervention Model Description: Interventional randomized placebo-controlled clinical trial. Adult, medullary injured (BM), with chronic neuropathic pain (DN). 4 groups: BM with DN with bedsore Ketamine Group versus Placebo Group BM with DN without bedsore group Ketamine versus Placebo Group Ketamine infusion 1 mg / kg IVSE over two hours versus Nacl perfusion 0.9%
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The randomisation is done with R software. Each randomisation card is put in a sealed opaque envelope. The two products being transparent, it's impossible to differentiate the two products with identical packaging is a syringe of 50 cc Luer Lock Plastipack BD with a standard extension for syringe Luer Lock.
  Both products will be prepared by an SSPI nurse who opens the envelope, the nurse does not participate in the study, the patient assessment investigator as well as the patient will remain blind about the administration of the product. Each syringe will be labeled for each patient with a special label without indication of the product The outcomes assessor, investigator and participant are blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Chronic neuropathic pain and bedsore Ketamine group (Active Comparator): Spinal cord injury population with central neuropathic pain at the lesional or sub-lesion level, chronically (for more than three months).
  Patients medullary wounded with chronic pain and ulcer pressure (inflammation factor).
  Midazolam 1mg before infusion. KETAMINE INFUSION IVSE 1mg/kg during 2 hours (0,5mg/kg/h). Preparation of 100mg in fifty cc, syringe with 2mg/ml. Rate of administration: Speed = Patient weight divided by four.
  Maximum 100mg. One and only perfusion.
  Interventions: Drug: Ketamine 10 MG/ML; Drug: Midazolam 1 MG/ML
- Chronic neuropathic pain and bedsore Placebo group (Placebo Comparator): Spinal cord injury population with central neuropathic pain at the lesional or sub-lesion level, chronically (for more than three months).
  Patients medullary wounded with chronic pain and ulcer pressure (inflammation factor).
  Midazolam 1mg before infusion. Sodium chloride infusion IVSE during 2 hours. Rate of administration : Speed = patient weight divided by four.
  One and only perfusion.
  Interventions: Drug: Placebos; Drug: Midazolam 1 MG/ML
- Chronic neuropathic pain without bedsore Ketamine group (Active Comparator): Spinal cord injury population with central neuropathic pain at the lesional or sub-lesion level, chronically (for more than three months).
  Patients medullary wounded with chronic pain and no ulcer pressure (no inflammation factor).
  Midazolam 1mg before infusion. KETAMINE INFUSION IVSE 1mg/kg during 2 hours (0,5mg/kg/h). Preparation of 100mg in fifty cc, syringe with 2mg/ml. Rate of administration: Speed = Patient weight divided by four.
  Maximum 100mg. One and only perfusion.
  Interventions: Drug: Ketamine 10 MG/ML; Drug: Midazolam 1 MG/ML
- Chronic neuropathic pain without bedsore Placebo group (Placebo Comparator): Spinal cord injury population with central neuropathic pain at the lesional or sub-lesion level, chronically (for more than three months).
  Patients medullary wounded with chronic pain and no ulcer pressure (no inflammation factor).
  Midazolam 1mg before infusion. Sodium chloride infusion IVSE during 2 hours. Rate of administration : Speed = patient weight divided by four.
  One and only perfusion.
  Interventions: Drug: Placebos; Drug: Midazolam 1 MG/ML

INTERVENTIONS:
Drug: Ketamine 10 MG/ML — Ketamine infusion 1mg/kg with electric syringe during 2 hours.
  Arms: Chronic neuropathic pain and bedsore Ketamine group; Chronic neuropathic pain without bedsore Ketamine group
Drug: Placebos — Sodium chloride infusion with the same rate, electric syringe during 2 hours.
  Other Names: Sodium chloride infusion
  Arms: Chronic neuropathic pain and bedsore Placebo group; Chronic neuropathic pain without bedsore Placebo group
Drug: Midazolam 1 MG/ML — Bolus of Midazolam 1mg before each perfusion.

SUMMARY:
The kynurenine pathway is involved in hyperalgesia. This pathway is activated by inflammation. Ketamine would interact with the kynurenine pathway and inflammation. Our working hypotheses are: the clinical effects of ketamine on neuropathic pain are greater in the presence of systemic inflammation and the mechanism of action involves an interaction on the kynurenine pathway.

Study design: Interventional randomized placebo-controlled clinical trial.

￼Main goals:

1. To show a better clinical efficacy of ketamine in chronic pain in patients with an inflammatory component.
2. Explore the anti-inflammatory activity of ketamine through the Kynurenine pathway.

DETAILED DESCRIPTION:
The kynurenine pathway is involved in hyperalgesia. This pathway is activated by inflammation. Ketamine would interact with the kynurenine pathway and inflammation. Our working hypotheses are: the clinical effects of ketamine on neuropathic pain are greater in the presence of systemic inflammation and the mechanism of action involves an interaction on the kynurenine pathway.

Study design: Interventional randomized placebo-controlled clinical trial.

￼Main goals:

1. To show a better clinical efficacy of ketamine in chronic pain in patients with an inflammatory component.
2. Explore the anti-inflammatory activity of ketamine through the Kynurenine pathway.

Population Adult, medullary injured (BM), with chronic neuropathic pain (DN). 4 groups: BM with DN with bedsore Ketamine Group versus Placebo Group BM with DN without bedsore group Ketamine versus Placebo Group

Intervention Ketamine infusion 1 mg / kg IVSE over two hours versus Nacl perfusion 0.9%

￼ Primary judgment criterion Decrease by more than 30% the intensity of neuropathic pain evaluated at the moment on a numerical scale of 10 points between H0 and H4. Comparison of groups two by two.

Secondary judgment criterions:

NPSI score (Neuropathic pain symptom inventory) at H1, H4, D1, D4, J7 Sub score of NPSI; H1, H4, J1, J4, J7 Depression Scale HADS (Hospital Anxiety Depression Scale) J0, J1, J7 Plasma serotonin (5-HT) kynurenine (KYN), indoleamine 2,3-dioxygenase 1 (IDO1) activity (KYN / TRP ratio), kynurenic acid ( KA) and quinolinic acid (QA), as well as 3 proinflammatory cytokines IL-1β, IL-6, and TNF-α before perfusion and H4 perfusion.

In parallel blood samples will be collected to study the activation of the kynurenine pathway in response to inflammation due to a pressure ulcer.

ELIGIBILITY:
Inclusion Criteria:

* Adults speaking and understanding French
* presenting chronic neuropathic pain as defined by IASP
* Painful intensity> or = to 6/10 during the week preceding the inclusion - Medullary lesion, whatever the origin (traumatic, degenerative, tumoral, postoperative), responsible for paraplegia in a chronic state.
* Able to give informed consent, after clear, fair and appropriate information
* Having given their consent by a written consent signature.

Exclusion Criteria:

* Hypersensitivity to ketamine or any of its components
* Participation in another interventional trial, or participation in another trial.
* Patient unable to give consent.
* Pregnancy or breastfeeding
* Refusal to sign the consent
* Cardiovascular diseases associated in particular with disorders of rhythm and severe cardiac insufficiency, coronary insufficiency, discovered on examination, on ECG or by biological balance or known. - unstabilized HTA> 180/100 mmHg
* Severe hepatic and / or renal hepatic insufficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2018-02-16 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Numeric pain rating scale decrease between H0 and H4. | 4 hours after the end of infusion
  Numeric pain rating scale is a scale from 0 to 10. 0 is no pain, 10 is the worst pain we could imagine. The first outcome is decreasing the intensity of neuropathic pain evaluated at the moment on a numerical scale of 10 points at H4. Comparison of groups two by two.

SECONDARY OUTCOMES:
Paraclinical: Kynurenine pathway levels : SEROTONIN | Hour 0 and Hour 6 (4 hours after the ending of infusion)
  Levels of SEROTONIN (millimoles/liter)
Paraclinical: Kynurenine pathway levels : KYNURENINE | Hour 0 and Hour 6 (4 hours after the ending of infusion)
  Levels of KYNURENINE (millimoles/liter)
Paraclinical: Kynurenine pathway levels : IDO ACTIVITY | Hour 0 and Hour 6 (4 hours after the ending of infusion)
  Levels of INDOLEAMINE DIOXYGENASE ACTIVITY (division Kynurenine/Tryptophane quote)
Paraclinical: Kynurenine pathway levels : KYNURENIC ACID | Hour 0 and Hour 6 (4 hours after the ending of infusion)
  Levels of Kynurenic acid (millimoles/liter)
Paraclinical: Kynurenine pathway levels : QUINOLINIC ACID | Hour 0 and Hour 6 (4 hours after the ending of infusion)
  Levels of Quinolinic acid (millimoles/liter)
Paraclinical: Kynurenine pathway levels : IL1 | Hour 0 and Hour 6 (4 hours after the ending of infusion)
  Levels of Interleukin 1 (picograms/milliliter)
Paraclinical: Kynurenine pathway levels : IL6 | Hour 0 and Hour 6 (4 hours after the ending of infusion)
  Levels of Interleukin 6 (picograms/milliliter)
Paraclinical: Kynurenine pathway levels: TNF alpha | Hour 0 and Hour 6 (4 hours after the ending of infusion)
  Levels of TNF alpha (picograms/milliliter)
Clinical: Neuropathic pain symptom inventory | Hour 0, Day 1, Day 4, Day 7
  NPSI scoring: Neuropathic pain symptom inventory. A composite score composed by neuropathic pain components: Burning, Pressure, Squeezing, Electric shocks, Stabbing, Evoked by brushing, evoked by pressure, evoked by cold stimuli, pins and needles, tingling. Two questions about the time of pain for twenty four hours, and the numbers of crisis. Score from 0 to 100. 100 is the maximum.
Clinical: Pain timeline | Seven days
  Timeline of self assessment on a simple numeric scale of the pain three times a day during a week. Numeric pain rating scale is a scale from 0 to 10. 0 is no pain, 10 is the worst pain we could imagine.
Percentage overall improvement in pain over a week with self assessment | Between Hour 0 and Day 7
  Self assessment of the global improvement in pain over the week after infusion
Clinical: Subscore of Neuropathic pain symptom inventory | Hour 0, Day 1, Day 4, Day 7
  Subscore on NPSI scoring: NEUROPATHIC PAIN SYMPTOM INVENTORY, subscore are burning from 0 to 10, pressing (deep) spontaneous pain from 0 to 10, paroxysmal pain from 0 to 10, evoked pain from 0 to 10, paresthesia or dysesthesia from 0 to 10 (0 is the minimal, 10 is the maximal value for each of the component).
Clinical: Hospital anxiety and depression scale | Hour 0, Day 7.
  Recording scoring on hospital anxiety and depression scale. HADS scale is a tool to detect anxiety and depressive disorders. It includes fourteen questions from 0 to 3 points each. Seven are related to anxiety. Seven are related to depressive mood. It permits to obtain 2 different scales with the maximum of each of 21.
Percentage overall improvement in mood over a week with self assessment | Between Hour 0 and day 7
  Self assessment of the global improvement of the mood over the week after infusion
Clinical: Pain area on a body cartography | Hour 0, Day 1, Day 7.
  Evaluation of pain area on a body surface cartography
Clinical: Ketamine adverse effects | Hour 0 to hour 4
  Recording ketamine adverse effects during and right after the infusion
Paraclinical: Kynurenine pathway activation with ulcer pressure | Hour 0
  Studying the levels of the kynurenine pathway elements between patients with inflammatory component (ulcer pressure) and without inflammatory component (without ulcer pressure)

CONTACTS AND LOCATIONS:
Overall Officials: Didier Bouhassira, Md, PhD, Study Chair — INSERM U987
Locations (1):
- Raymond Poincaré Hospital, Garches, Hauts De Seine, France

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-30): https://cdn.clinicaltrials.gov/large-docs/22/NCT03513822/Prot_SAP_000.pdf